CLINICAL TRIAL: NCT05092373
Title: Phase I Study of Tumor Treating Fields (TTF) in Combination With Cabozantinib or With Pembrolizumab and Nab-Paclitaxel in Patients With Advanced Solid Tumors Involving the Abdomen or Thorax
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0299; NCI-2021-11360 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0299 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Carcinoma; Advanced Endometrial Carcinoma; Advanced Fallopian Tube Carcinoma; Advanced Hepatocellular Carcinoma; Advanced Malignant Abdominal Neoplasm; Advanced Malignant Female Reproductive System Neoplasm; Advanced Malignant Thoracic Neoplasm; Advanced Ovarian Carcinoma; Advanced Primary Peritoneal Carcinoma; Advanced Renal Cell Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Malignant Abdominal Neoplasm; Malignant Solid Neoplasm; Metastatic Breast Carcinoma; Metastatic Endometrial Carcinoma; Metastatic Fallopian Tube Carcinoma; Metastatic Hepatocellular Carcinoma; Metastatic Malignant Abdominal Neoplasm; Metastatic Malignant Female Reproductive System Neoplasm; Metastatic Malignant Thoracic Neoplasm; Metastatic Ovarian Carcinoma; Metastatic Primary Peritoneal Carcinoma; Metastatic Renal Cell Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Stage III Fallopian Tube Cancer AJCC v8; Stage III Hepatocellular Carcinoma AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage III Uterine Corpus Cancer AJCC v8; Stage IIIA Fallopian Tube Cancer AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Primary Peritoneal Cancer AJCC v8; Stage IIIA Uterine Corpus Cancer AJCC v8; Stage IIIA1 Fallopian Tube Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Fallopian Tube Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Fallopian Tube Cancer AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Primary Peritoneal Cancer AJCC v8; Stage IIIB Uterine Corpus Cancer AJCC v8; Stage IIIC Fallopian Tube Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Primary Peritoneal Cancer AJCC v8; Stage IIIC Uterine Corpus Cancer AJCC v8; Stage IIIC1 Uterine Corpus Cancer AJCC v8; Stage IIIC2 Uterine Corpus Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Hepatocellular; Ovarian Neoplasms; Carcinoma, Renal Cell | interventions — atezolizumab; cabozantinib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Cohort 1 (TTF, cabozantinib) (Experimental): Patients receive TTF continuously for at least 18 hours per day on days 1-21 of each cycle. Patients also receive cabozantinib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Procedure: Tumor Treating Fields Therapy
- Cohort 2 (TFF, atezolizumab, nab-paclitaxel) (Experimental): Patients receive TTF continuously for at least 18 hours per day on days 1-28 of each cycle. Patients also receive nab-paclitaxel IV over 30 minutes on days 1, 8, and 15 of each cycle and atezolizumab IV over 30-60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Nab-paclitaxel; Procedure: Tumor Treating Fields Therapy

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
  Arms: Cohort 2 (TFF, atezolizumab, nab-paclitaxel)
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184
  Arms: Cohort 1 (TTF, cabozantinib)
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
  Arms: Cohort 2 (TFF, atezolizumab, nab-paclitaxel)
Procedure: Tumor Treating Fields Therapy — Receive TTF
  Other Names: Alternating Electric Field Therapy; TTF; TTFields

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of tumor treating fields therapy in combination with either cabozantinib or nab-paclitaxel and atezolizumab in treating patients with solid tumors involving the abdomen or thorax that have spread to other parts of the body (advanced). Tumor treating fields therapy on this study utilizes NovoTTF systems that are wearable devices that use electrical fields at different frequencies that may help stop the growth of tumor cells by interrupting cancer cells' ability to divide. Cabozantinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals tumor cells to multiply. This helps slow or stop the spread of tumor cells. Chemotherapy drugs, such as nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving tumor treating fields therapy in combination with either cabozantinib, or with nab-paclitaxel and atezolizumab may help control advanced solid tumors involving the abdomen or thorax.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and tolerability of TTF, including the maximum tolerated dose (MTD), in combination with cabozantinib (Cohort 1) with nab-paclitaxel and pembrolizumab (Cohort 2) in patients with advanced solid tumors involving the abdomen or thorax to the 4 prespecified tumor types.

SECONDARY OBJECTIVE:

I. To assess the objective response rate, progression-free survival and overall survival of TTF in combination with cabozantinib (Cohort 1) with nab-paclitaxel and pembrolizumab (Cohort 2) in patients with advanced solid tumors involving the abdomen or thorax to the 4 prespecified tumor types.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients receive TTF continuously for at least 18 hours per day on days 1-21 of each cycle. Patients also receive cabozantinib orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

COHORT 2: Patients receive TTF continuously for at least 18 hours per day on days 1-28 of each cycle. Patients also receive nab-paclitaxel intravenously (IV) over 30 minutes on days 1, 8, and 15 of each cycle and atezolizumab IV over 30-60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed advanced/metastatic solid cancer (hepatocellular carcinoma, renal cell carcinoma, breast cancer, ovarian/fallopian, or endometrial/primary peritoneal tumors) involving the abdomen or thorax, cannot tolerate standard therapy or have experienced tumor progression on standard therapy.
* Age: ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy >3 months.
* Normal bone marrow function, defined as absolute neutrophil count ≥1,000/µL; platelets ≥75,000/µL; hemoglobin ≥8 g/dL.
* Adequate hepatic function as defined by a total bilirubin level ≤1.5 x the upper limit of normal (ULN), unless the patient has known Gilbert's syndrome, and alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase levels (SGPT) ≤2.5 x ULN (unless the patient has liver metastases: ALT)/ serum glutamic pyruvic transaminase levels (SGPT) ≤5 x ULN).
* Participants with HCC must have a Child Pugh status A, no clinically significant ascites (requiring pharmacological or interventional treatment), and no history (or increased risk) of esophageal/gastric bleeding, impaired wound healing, perforation or fistula.
* Serum creatinine clearance ≥50 mL/min by the Cockcroft-Gault formula.
* Measurable disease by RECIST or evaluable disease.
* Contraception: Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months and who have not had a tubal ligation, hysterectomy, or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately. Male participants must agree to use effective contraception or abstinence while on study.
* Able to operate the TTF device independently or with the help of a caregiver.

Exclusion Criteria:

* Participants must not receive prior anticancer therapy or radiation therapy within 2 weeks and must not undergo major surgery within 4 weeks prior to initiation of treatment on protocol. Participants who are already on cabozantinib and have progressive disease are allowed to transition to treatment with tumor treating fields and cabozantinib. Participants in both cohorts who already started treatments as standard of care (Cohort 1: Cabozantinib and Cohort 2: nab-paclitaxel and Pembrolizumab) are allowed to start on protocol within the first 2-3 weeks of treatment initiation. Palliative radiation therapy is allowed.
* Participants must have recovered to Grade 0-1 toxicity from prior therapy.
* Active brain metastasis or leptomeningeal disease. Patients with treated brain metastasis must have stable disease, evidenced by brain imaging for at least 4 weeks and the patient must have been off steroids for at least 2 weeks.
* The patient has cardiac conditions as follows: uncontrolled: hypertension (blood pressure [BP] > 160/100) despite optimal therapy, uncontrolled angina, ventricular arrhythmias, congestive heart failure (New York Heart Association Class II or above), prior or current cardiomyopathy, uncontrolled atrial fibrillation with heart rate > 100 beats per minute (bpm), unstable ischemic heart disease (myocardial infarction within 6 months prior to starting treatment or angina requiring use of nitrates more than once weekly).
* The patient has concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes, severe infection requiring active treatment, severe malnutrition, chronic severe liver or renal disease).
* Concurrent malignancies are permitted if (A) they were previously treated, and all treatment of that malignancy was completed at least 2 years before enrollment and no evidence of disease exists, or (B) with agreement from the Principal Investigator (PI), participants who have a concurrent malignancy that is clinically stable and does not require tumor-directed treatment are eligible to participate if the risk of the prior malignancy interfering with either safety or efficacy endpoints is very low, or (C) with agreement from the PI, other malignancies may be permitted if the risk of the prior malignancy interfering with either safety or efficacy end points is very low. Adequately treated basal or squamous cell carcinoma or carcinoma in situ is allowed.
* The patient is pregnant or breastfeeding.
* History of hypersensitivity or contraindication to TTF.
* Implanted pacemaker, defibrillator or other electrical medical devices.
* The participant has a previously-identified allergy or hypersensitivity to cabozantinib, nab-paclitaxel, or pembrolizumab, medical adhesives or hydrogel or the patient has received prior cabozantinib and discontinued therapy due to unacceptable toxicity.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* The patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* CABOZANTINIB COHORT ONLY: The patient has experienced clinically-significant hematemesis or hemoptysis of > 0.5 teaspoon of red blood, or other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment.
* CABOZANTINIB COHORT ONLY: The patient has a cavitating pulmonary lesion(s) or a pulmonary lesion abutting or encasing a major blood vessel.
* CABOZANTINIB COHORT ONLY: The patient has received drugs used to control loss of bone mass within 4 weeks prior to the first dose of study treatment.
* CABOZANTINIB COHORT ONLY: The patient has prothrombin time/international normalized ratio (PT/INR) or partial thromboplastin time (PTT) test results that are above (1.3X) the laboratory upper limit of normal.
* CABOZANTINIB COHORT ONLY: The subject has a corrected QT interval (QTcF) > 450 ms for men or > 470 ms for women.
* CABOZANTINIB COHORT ONLY: The patient requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or Coumadin-related agents, heparin, thrombin or FXa inhibitors, and antiplatelet agents. Low-dose aspirin (≤ 81 mg/day), low dose warfarin (≤ 1mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted.
* CABOZANTINIB COHORT ONLY: Patients with encasement of a major artery or bowel by tumor are excluded.
* CABOZANTINIB COHORT ONLY: The patient is unable to swallow capsules.
* CABOZANTINIB COHORT ONLY: History of hypersensitivity or contraindication to cabozantinib.
* ATEZOLIZUMAB-CONTAINING COHORT: Participants who have received prior immunotherapy, including prior anti-PD-1 or anti-PD-L1 therapies may participate: (A) only if their prior anti-PD-1 or anti-PDL1 monotherapy or combination therapy were NOT the last treatment prior to participation on this study. (B) Participants who had prior immunotherapies and experienced Grade 1-2 immune-related adverse event (irAE) must have documentation that their irAEs are Grade 1 or 0 using current Common Terminology Criteria for Adverse Events v5.0 (CTCAE v5.0) and participants must be off steroid therapy and/or other immunosuppressive therapy, as treatment for irAEs, for >= 14 days from Cycle 1, Day 1. (C) Participants who experienced Grade 3 irAEs consisting of laboratory abnormalities that were asymptomatic and have now resolved to Grade 1 or 0 and participants who have been off steroid and/or other immunosuppressive therapy, as treatment for irAEs, for >= 30 days from Cycle 1, Day 1. Participants with prior irAE pneumonitis (>= Grade 2) should not be given atezolizumab.
* ATEZOLIZUMAB-CONTAINING COHORT: Human immunodeficiency virus (HIV) infection, active Hepatitis B or C infection, or active infections requiring oral or intravenous antibiotics.
* ATEZOLIZUMAB-CONTAINING COHORT: Has received a live vaccine within 30 days prior to first dose.
* ATEZOLIZUMAB-CONTAINING COHORT: Active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation.
* ATEZOLIZUMAB-CONTAINING COHORT: Serious autoimmune disease at the discretion of the treating attending: Patients with a history of active serious inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus or autoimmune vasculitis (e.g. Wegener's Granulomatosis) are excluded from this study.
* ATEZOLIZUMAB-CONTAINING COHORT: History of/or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of TTF, including the maximum tolerated dose (MTD). | through study completion, an average of 2 to 3 years
  To assess the safety and tolerability of TTF, including the maximum tolerated dose (MTD),in combination with cabozantinib (Cohort 1) or with nab-paclitaxel and atezolizumab (Cohort 2) in patients with advanced solid tumors involving the abdomen or thorax to the 4 prespecified tumor types. 1st cycle with at least 6 evaluable patients treated at the dose.

SECONDARY OUTCOMES:
To assess the objective response rate, progression-free survival and overall survival | through study completion, an average of 2 to 3 years
  To assess the objective response rate, progression-free survival and overall survival of TTF in combination with cabozantinib (Cohort 1) or with nab-paclitaxel and atezolizumab (Cohort 2) in patients with advanced solid tumors involving the abdomen or thorax to the 4 prespecified tumor types.sion 1.1. Will be estimated along with its exact 95% confidence interval (CI). Patients who were replaced without tumor evaluation will not be included in ORR estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M Tsimberidou, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org